CLINICAL TRIAL: NCT04704245
Title: A Randomized Controlled Trial on the Effectiveness of Epidermal Growth Factor-containing Ointment on the Treatment of Solar Lentigines as Adjuvant Therapy
Brief Title: Effectiveness of Epidermal Growth Factor-containing Ointment on the Solar Lentigines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Bo Young Chung, Principal Investigator, Clinical Professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-06-009
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Epidermal Growth Factor; Nd-yttrium Aluminum Garnet Laser; Hyperpigmentation; Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation | interventions — Epidermal Growth Factor; Long-Term Synaptic Depression; Lasers; BRCA1 Protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epidermal growth factor (EGF) containing ointment group (Experimental): The subjects received one session of laser treatment with a Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser after enrollment.
  The procedure parameters were as follows: 5-10-ns pulse duration, 3.5-mm spot size, 0.9-1.1-J/cm2 fluence, and 2-Hz frequency.
  The end point of laser treatment for lentigines was immediate whitening. The subjects then applied the epidermal growth factor (EGF) ointment twice daily (morning and evening) to the lesion for 4 weeks after laser treatment.
  Interventions: Drug: epidermal growth factor (EGF)-containing ointment; Procedure: Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser
- Vehicle ointment group (Placebo Comparator): The subjects received one session of laser treatment with a Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser of their solar lentigines after enrollment.
  The procedure parameters were as follows: 5-10-ns pulse duration, 3.5-mm spot size, 0.9-1.1-J/cm2 fluence, and 2-Hz frequency.
  The end point of laser treatment for lentigines was immediate whitening. The subjects then applied the vehicle ointment twice daily (morning and evening) to the lesion for 4 weeks after laser treatment.
  Interventions: Drug: Vehicle ointment; Procedure: Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser

INTERVENTIONS:
Drug: epidermal growth factor (EGF)-containing ointment — The subjects applied the epidermal growth factor (EGF) ointment twice daily (morning and evening) to the lesion for 4 weeks after laser treatment.
  Other Names: Easyef Saesal ointment, Daewoong Pharmaceutical Co., Ltd., Seoul, Korea
  Arms: epidermal growth factor (EGF) containing ointment group
Drug: Vehicle ointment — To compare the effect of epidermal growth factor (EGF) ointment, the control subjects applied the vehicle ointment twice daily (morning and evening) to the lesion for 4 weeks after laser treatment.
  Other Names: containing petrolatum
  Arms: Vehicle ointment group
Procedure: Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser — The subjects received one session of laser treatment with a Q-swithced (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser of their solar lentigines after enrollment.
  The procedure parameters were as follows: 5-10-ns pulse duration, 3.5-mm spot size, 0.9-1.1-J/cm2 fluence, and 2-Hz frequency.
  The end point of laser treatment for lentigines was immediate whitening.
  Other Names: Nd:yttrium aluminum garnet laser (Iris, Bluecore Company Co., Ltd., Busan, Korea)

SUMMARY:
Subjects were randomly assigned to groups for treatment with either an EGF-containing ointment (the study group) or the vehicle alone (petrolatum; the control group). The EGF ointment included recombinant human EGF (1 μg/g). Random numbers used for assignment to groups were provided by the randomization function of SAS.

The subjects received one session of laser treatment with a Q-switched (QS) 532-nm Nd:yttrium aluminum garnet (YAG) laser of their solar lentigines after enrollment. . The end point of laser treatment for lentigines was immediate whitening. The subjects then applied the EGF ointment or vehicle twice daily (morning and evening) to the lesion for 4 weeks after laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of solar lentigines that occurred after adulthood
* age of 20 years or older.

Exclusion Criteria:

* uncontrolled systemic or chronic disease
* hypersensitivity to the ingredients of the ointment
* current use of skin whitening agents
* a history of other laser treatments within the past 6 months
* pregnancy
* lactation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Change of pigmentation by physician's assessment | Change from baseline pigmentation at 4 weeks
  The pigment clearance was assessed using a 5-grade percentage improvement scale
  grade 1, <0% [worse]; grade 2, 0%-25% improvement; grade 3, 26%-50% improvement; grade 4, 51%-75% improvement; grade 5, 76%-100% improvement
  -> higher score means better outcomes
Change of pigmentation by physician's assessment | Change from baseline pigmentation at 8 weeks
  The pigment clearance was assessed using a 5-grade percentage improvement scale
  grade 1, <0% [worse]; grade 2, 0%-25% improvement; grade 3, 26%-50% improvement; grade 4, 51%-75% improvement; grade 5, 76%-100% improvement
  -> higher score means better outcomes

SECONDARY OUTCOMES:
Erythema index | baseline
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine erythema.
Erythema index | 2 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine erythema.
Erythema index | 4 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine erythema.
Erythema index | 8 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine erythema.
Melanin index | baseline
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine pigmentation.
Melanin index | 2 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine pigmentation.
Melanin index | 4 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine pigmentation.
Melanin index | 8 weeks
  A spectrophotometer was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine pigmentation.
Transepidermal water loss | baseline
  A VapoMeter®(Delfin Technologies Ltd., Kuopio, Finland) was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine transepidermal water loss
Transepidermal water loss | 2 weeks
  A VapoMeter®(Delfin Technologies Ltd., Kuopio, Finland) was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine transepidermal water loss
Transepidermal water loss | 4 weeks
  A VapoMeter®(Delfin Technologies Ltd., Kuopio, Finland) was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine transepidermal water loss
Transepidermal water loss | 8 weeks
  A VapoMeter®(Delfin Technologies Ltd., Kuopio, Finland) was used to assess the lesion in a room at constant temperature (20-24 °C) and humidity (28%-38%).
  Skin measurements were performed to determine transepidermal water loss
Patient's subjective satisfaction | 4 weeks
  The patient's subjective satisfaction was assessed by questionnaire according to the following: 1, worse; 2, no change; 3, mild improvement; 4, moderate improvement; or 5, significant improvement.
  higher score means better outcome
Patient's subjective satisfaction | 8 weeks
  The patient's subjective satisfaction was assessed by questionnaire according to the following: 1, worse; 2, no change; 3, mild improvement; 4, moderate improvement; or 5, significant improvement.
  higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Chung, M.D., PhD, Study Chair — Department of Dermatology, Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HO, Kim HR, Kim JC, Kang SY, Jung MJ, Chang SE, Park CW, Chung BY. A Randomized Controlled Trial on the Effectiveness of Epidermal Growth Factor-Containing Ointment on the Treatment of Solar Lentigines as Adjuvant Therapy. Medicina (Kaunas). 2021 Feb 13;57(2):166. doi: 10.3390/medicina57020166. PMID 33668564